CLINICAL TRIAL: NCT05859841
Title: Effect of Music Listening at Acute Stage of Stroke on the Recovery and Quality of Life: Block-randomized Controlled Study
Brief Title: Effect of Music Listening on Stress in Acute Stroke
Acronym: MUKU3-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Seppo Soinila, Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34/1801/2017
Record Dates: First submitted 2017-06-09; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Stroke
Keywords: Stroke; Music; stress
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: 15 pt listen to music, 15 receives standard treatment, care and rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music listening (Experimental): Music listening under instruction by music therapist, min 3 hours daily
  Interventions: Other: Music listening
- Control (Placebo Comparator): Standard treatment, care and rehabilitation
  Interventions: Other: Control

INTERVENTIONS:
Other: Music listening — Music listening under instruction by music therapist, min 3 hours daily
  Arms: Music listening
Other: Control — Standard treatment, care and rehabilitation
  Arms: Control

SUMMARY:
Investigation on changes in the neurochemical stress parameters in acute stroke. 30 patients are recruited in the stroke unit, blood samples are collected at fixed intervals during the first two days. Patients are randomized to music listening and control.Neuropsychological testing is performed in the acute phase and 6 months post-stroke.

DETAILED DESCRIPTION:
Outcome measures: NIHSS, stress hormone levels, questionnaires on mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hemispheric infarction
* Neurologically stable

Exclusion Criteria:

* Previous neurological disease affecting the outcome
* Previous psychiatric disease affecting the outcome
* Substance abuse

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale | 1 day post-stroke
  Change in Depression, Anxiety and Stress Scale scores
National Institute of Health Stroke Scale | 1 day post-stroke
  Change in National Institute of Health Stroke Scale scores
Visual Analogue Mood Scale | 2 days post stroke
  Change in Visual Analogue Mood Scale scores
Serum cortisol | 2 days post-stroke
  Change in serum cortisol level
Serum C-reactive protein | 2 days post-stroke
  Change in serum C-reactive protein level
Montreal Cognitive Assessment | 3 days post-stroke
  Montreal Cognitive Assessment score
Blood pressure | 3 days post-stroke
  Change in systolic/diastolic blood pressure
Pulse rate | 3 days post-stroke
  Change in pulse rate
Depression, Anxiety and Stress Scale | 6 months post-stroke
  Change in Depression, Anxiety and Stress Scale scores
National Institute of Health Stroke Scale | 6 months post-stroke
  Change in National Institute of Health Stroke Scale
Visual Analogue Mood Scale | 6 months post-stroke
  Change in Visual Analogue Mood Scale scores
Montreal Cognition Assessment | 6 moths post-stroke
  Change in Montreal Cognition Assessment score
Stroke and Aphasia Quality of Life scale | 6 months post-stroke
  Change in Stroke and Aphasia Quality of Life scale score
Center for Epidemiological Studies Depression score | 6 months post-stroke
  Change in Center for Epidemiological Studies Depression score
Working Memory Questionnaire | 6 months post-stroke
  Change in Working Memory Questionnaire score
Stroke Impact Scale | 6 months post-stroke
  Change in Stroke Impact Scale score

SECONDARY OUTCOMES:
Leisure Activity Questionnaire | 6 months post-stroke
  Change in leisure activities (pre- vs. post-stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Tuomaala, Study Chair — Chief of Research
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No